CLINICAL TRIAL: NCT01587469
Title: Evaluation of Xpert MTB/RIF Assay for the Rapid Identification of TB and TB Rifampin Resistance in HIV-Infected and HIV-Uninfected Pulmonary Tuberculosis Suspects
Brief Title: Evaluation of Xpert MTB/RIF Assay for the Rapid Identification of TB and TB Rifampin Resistance in Pulmonary Tuberculosis Suspects
Status: Completed | Type: Observational
Sponsor: Cepheid (Industry)
Collaborators: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: ACTG A5295
Record Dates: First submitted 2012-04-24; First posted 2012-04-30 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Samples of sputum may be retained

GROUPS / COHORTS (1):
- HIV-infected and -uninfected individuals: HIV-infected and -uninfected individuals with suspected TB infection

SUMMARY:
This observational Mycobacterium tuberculosis (MTB) diagnostics evaluation study is a longitudinal study of pulmonary TB suspects who are undergoing sputum evaluation for pulmonary TB. The sensitivity and specificity of the Xpert MTB/RIF (Mycobacterium tuberculosis/rifampin) assay performed on the first sputum collected for Xpert testing will be compared to gold standard conventional culture methods on two sputum specimens, in HIV-infected and HIV-uninfected participants.

ELIGIBILITY:
Inclusion Criteria:

* Suspected pulmonary TB (more information on the criterion can be found in the protocol)
* Men and women age equal to or greater than 18 years
* Ability and willingness of candidate or legal guardian/representative to provide informed consent
* Collection of two sputum samples for AFB smear and culture collected within 7 days prior to entry.
* Availability of two samples for Xpert MTB/RIF testing collected within 7 days prior to entry.
* Determination and/or documentation of HIV status
* For HIV-positive candidates, a CD4+ cell count obtained within 45 days prior to study entry or drawn at the time of entry at any laboratory that has a CLIA certification or its equivalent.

Exclusion Criteria:

* Either receipt of ≥48 cumulative hours OR three or more doses of anti-TB treatment within 180 days prior to completion of second sputum collection for Xpert testing
* Receipt of more than 7 cumulative days of antibiotics intended for bacterial treatment that may have anti-tuberculosis activity, within the 14 days prior to first sputum collection
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-1-infected and -uninfected men and women, 18 years and older, pulmonary TB suspects who have either a) smear positive sputum or b) clinical suspicion of pulmonary TB including one or more self-reported symptoms of cough, night sweats, weight loss, or fever. Within the 180 days prior to collection of the initial sputum sample, participants will have received none or fewer than 48 hours of TB treatment and, in those 48 hours, fewer than three doses of TB treatment.
Sampling Method: Non-Probability Sample
Enrollment: 992 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2014-02-21 (Actual); Study Completion 2014-02-21 (Actual)

PRIMARY OUTCOMES:
Proportion of all participants with Xpert MTB/RIF Assay MTB positive in sputum #1 who are AFB smear positive and MGIT culture positive for M.tuberculosis. | Week 0
Proportion of all participants with Xpert MTB/RIF Assay MTB positive in sputum #1 who are AFB smear negative and MGIT culture positive for M.tuberculosis. | Week 0
Proportion of US participants with Xpert MTB/RIF Assay MTB negative in sputum #1 who are MGIT culture negative for M.tuberculosis. | Week 0

CONTACTS AND LOCATIONS:
Overall Officials: Annie Luetkemeyer, MD, Study Chair — San Francisco General Hospital; Cynthia Firnhaber, MD, Study Chair — University of Witwatersrand, South Africa
Locations (1):
- Ucsf Aids Ctu, San Francisco, California, United States

REFERENCES:
- [Result] Luetkemeyer AF, Firnhaber C, Kendall MA, Wu X, Mazurek GH, Benator DA, Arduino R, Fernandez M, Guy E, Johnson P, Metchock B, Sattler F, Telzak E, Wang YF, Weiner M, Swindells S, Sanne IM, Havlir DV, Grinsztejn B, Alland D; AIDS Clinical Trials Group A5295 and Tuberculosis Trials Consortium Study 34 Teams. Evaluation of Xpert MTB/RIF Versus AFB Smear and Culture to Identify Pulmonary Tuberculosis in Patients With Suspected Tuberculosis From Low and Higher Prevalence Settings. Clin Infect Dis. 2016 May 1;62(9):1081-8. doi: 10.1093/cid/ciw035. Epub 2016 Feb 2. PMID 26839383